CLINICAL TRIAL: NCT04013919
Title: Observational, Data Collection Study for Subjects With Diabetes Using Daily Insulin Injections and Monitoring Glucose by Continuous Glucose Monitoring or Self-Monitoring Blood Glucose
Brief Title: Observational, Data Collection Study for Subjects With Diabetes Using Insulin Injections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DreaMed Diabetes (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-0999
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 Diabetes
  Interventions: Drug: Multiple Daily Injections of Insulin
- Type 2 Diabetes
  Interventions: Drug: Multiple Daily Injections of Insulin; Drug: Single insulin injections

INTERVENTIONS:
Drug: Multiple Daily Injections of Insulin — Basal/ Bolus insulin injections
Drug: Single insulin injections — Basal insulin injections only
  Groups: Type 2 Diabetes

SUMMARY:
This is an observational, multicenter prospective study including up to 260 subjects with type 1 or type 2 diabetes who use insulin injections (either basal insulin only or multiple daily injections (MDI)) and CGM or SMBG to manage their diabetes. The study aims to generate the database needed for future development and verification of insulin-glucose modules of subjects with diabetes using insulin injections.

During the study, subjects will continue their regular diabetes management using their regular glucose monitoring method (either CGM or SMBG), insulin injections and oral medication (as applicable). Subjects will be requested to document glucose levels and insulin delivery during basal only or basal/bolus insulin treatment. In addition, subjects will have their daily activities recorded (meals, physical activity etc) using electronic log (implemented on the CGM/FGM receiver, Dedicated App, Neura App and/or other logbooks). Data will be captured during regular daily life using Insulin Connected pens and daily diary application software, for a period of 1 month.

ELIGIBILITY:
Inclusion Criteria:

1. Documented T1D or T2D for at least 1 year prior to study enrolment
2. T1D: Subjects aged 1 year or older
3. T2D: Subjects aged 30 years or older
4. A1c at inclusion ≤ 10%
5. Subjects using basal-bolus MDI therapy or basal insulin only - basal insulin Lantus or Tregludec and any short acting insulin.

   * T2D: Insulin pumps will also be accepted.
6. T2D: BMI ≥ 25 kg/m2
7. Subjects willing to follow study instructions:

   1. For SMBG users: measure capillary blood glucose at least 4 times a day and twice a week 7-point profile. Document blood glucose level, insulin delivery, meals and daily activities. Optional: wear blinded CGM.
   2. For CGM users: Document insulin delivery, meals and daily activities. Optional:

   Measure capillary blood glucose in addition.
8. Adult subjects or parents of pediatric subjects willing and able to sign a written informed consent form.

Exclusion Criteria:

1. An episode of diabetic keto-acidosis within the month prior to study entry and/or severe hypoglycemia resulting in seizure or loss of consciousness in the month prior to enrolment.
2. Concomitant diseases/ treatment that influence metabolic control (except diabetes treatment for T2) or any significant diseases /conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study or compromise subject's safety
3. T2D: eGFR < 60
4. Participation in any other interventional study
5. Female subject who is pregnant or planning to become pregnant within the planned study duration
6. T1D: Subject is in the "honeymoon" phase - i.e. less than 0.5 insulin units/kg per day.
7. Drug or alcohol abuse.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 260 subjects with diabetes mellitus will be recruited in the following distribution: up to 100 T1D and up to 160 T2D. All subjects will be using multiple daily injections of insulin or basal injections only and self-monitoring blood glucose or continuous glucose monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Glucose levels | 1 month
  Characterise the insulin-glucose dynamics for insulin users

CONTACTS AND LOCATIONS:
Locations (1):
- Scheider MC, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No